CLINICAL TRIAL: NCT00505518
Title: Feasibility and Effectiveness of Telepsychiatry for Collaborative Management of Chinese Americans With Psychiatric Disorders in a Nursing Home
Brief Title: Investigating the Effectiveness of Telepsychiatry for Treating Major Depression in a Chinese American Nursing Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Albert Yeung, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-P-001508
Record Dates: First submitted 2007-07-19; First posted 2007-07-23 (Estimated); Results first posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-07

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Telepsychiatry; Chinese American; Nursing Home
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Psychotropic medication (at discretion of psychiatrist) — Antidepressant medication, prescribed at discretion of psychiatrist
Behavioral: Collaborative psychiatric and primary medical care — Regular care visits from health workers

SUMMARY:
The current use of telepsychiatry, or psychiatric care using videoconferencing, is very limited. The present study investigates the use of this method with a depressed Chinese American population in a nursing home. It is believed that this population can benefit from telepsychiatric treatment when used in collaboration with the primary care they receive in the nursing home.

DETAILED DESCRIPTION:
Individuals at the South Cove Manor nursing home will be referred to this study if they are experiencing depression. After meeting with the Principal Investigator (a psychiatrist), he will collaborate with the primary care physician and the nursing home staff to establish a treatment plan for the patient. Videoconferencing will be used by the P.I. for regular psychiatric visits with the patient as well as meetings with the nursing home staff to coordinate care for the patient. After collaboration between the two groups, treatment suggestions will be given to the patient's primary care physician (PCP) to implement in the primary care setting. The patient's symptomology, mood, satisfaction of life and side effects of medication will be recorded regularly to measure the effects of treatment for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Major Depressive Disorder
* Patient at South Cove Manor Nursing Home
* Referred by nursing staff for psychiatric consultation

Exclusion Criteria:

* Not competent to participate in psychiatric interviews

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Yeung, S., M.D., Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Depression and Clinical Research Program at Massachusetts General Hospital, Boston, Massachusetts
  - South Cove Manor, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from September 2006 to November 2007 as a collaborative project between Massachusetts General Hospital and South Cove Manor Nursing Home, which is located in Boston's Chinatown.
Groups:
- Telepsychiatry Treatment: Patients in the telepsychiatry treatment group will videoconference the P.I. for regular psychiatric visits in addition to meeting with nursing home staff. Treatment suggestions will be provided to the patient's primary care physician to be implemented.
Period: Overall Study
Arm/Group | Telepsychiatry Treatment
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Telepsychiatry Treatment
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 77.33 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Scores on Clinical Global Impressions
Description: Minimum score - 1 (better outcome) Maximum score - 7 (worse outcome)
Time Frame: Baseline, 30 days or 60 days (length depended on clinical needs of patients)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Telepsychiatry: Telepsychiatry-based follow up visits with psychiatrist.
Arm/Group | Telepsychiatry
Number analyzed (Participants) | 9
units on a scale | -2.1 (0.38)

2. Primary Outcome: Patient/Family Telepsychiatry Service Satisfaction Survey
Description: Patients' (or their family members' for those who had severe cognitive deficits) satisfaction with the telepsychiatry services were surveyed using a satisfaction questionnaire specifically designed for this study. The satisfaction questionnaire is a scale with three choices: "not satisfied", "satisfied", and "highly satisfied."
Time Frame: 30 days or 60 days (length depended on clinical needs of patients)
Measure: Number; unit: participants
Arm/Group | Telepsychiatry
Number analyzed (Participants) | 9
participants
  Highly not satisfied | 0
  Not satisfied | 0
  Satisfied | 1
  Highly satisfied | 7
  No response | 1

3. Primary Outcome: Nurse Telepsychiatry Services Satisfaction Questionnaire
Description: The charge nurse's satisfaction with the telepsychiatry services were surveyed using a satisfaction questionnaire specifically designed for this study. The satisfaction questionnaire is a scale with three choices: "not satisfied", "satisfied", and "highly satisfied."
Time Frame: 30 days or 60 days (length depended on clinical needs of patients)
Measure: Number; unit: Participants
Arm/Group | Telepsychiatry
Number analyzed (Participants) | 9
Participants
  Highly Satisfied | 8
  Satisfied | 1
  Not Satisfied | 0

ADVERSE EVENTS:
Arm/Group | Telepsychiatry Treatment
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
Many subjects in the study suffered from dementia and psychotic symptoms, thus their responses may not be reliable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes